CLINICAL TRIAL: NCT00562341
Title: Effect of Lap-Band Induced Weight Loss on Serum PSA Levels, Testosterone, Estrogen and Other Serum Markers
Brief Title: Effect of Lap-Band Induced Weight Loss on Serum PSA Levels
Status: Withdrawn | Type: Observational
Why Stopped: enrollment challenges
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 07/09/VA18
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Obesity; Prostate Cancer
Keywords: obesity; psa; prostate cancer
MeSH Terms: conditions — Obesity; Prostatic Neoplasms; Salivary Gland Adenoma, Pleomorphic | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- bariatric surgery: description of enrollees
  Interventions: Other: Bariatric Surgery

INTERVENTIONS:
Other: Bariatric Surgery — one time lapb-band gastric bypass surgery

SUMMARY:
The proposed prospective study aims to determine whether interpretation of PSA levels in morbidly obese men require correction due to the obesity itself. If PSA levels are found to rise after weight loss, interpretation of PSA levels in morbidly obese men may be improved by upward correction of the PSA level. A 'correction factor' may be proposed for the interpretation of PSA levels in obese men, toward the clinical decision regarding indication for prostate biopsy.

DETAILED DESCRIPTION:
The main objective of this study is to determine whether interpretation of PSA levels in morbidly obese men require correction due to the obesity itself. Secondary outcome measures that will be followed include the affect of obesity and weight loss on testosterone, estradiol and leptin. In as much as these might also affect PSA, we will be measuring these values as well. Also, we do not know the effects of lap-band induced weight loss on clinical outcome measures of sexual, bowel and urinary function. Thus we will aim to investigate these parameters as well.

ELIGIBILITY:
Inclusion Criteria:

* obese men undergoing lap-band surgery

Exclusion Criteria:

* prior diagnosis of prostate cancer
* prior prostate surgery
* use of 5-alpha reductase inhibitors
* history of prostatitis
* recurrent Urinary Tract Infection (UTI).

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients asked to enroll will be obese men who are undergoing bariatric surgery, lap-band surgery, at Maimonides Medical Center.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12-31 (Actual); Study Completion 2009-12-31 (Actual)

PRIMARY OUTCOMES:
Prostate-Specific Antigen (PSA) value | 18 months
  The PSA serum test measures the level of PSA in a man's blood. The results are usually reported as nanograms of PSA per milliliter (ng/mL) of blood.

SECONDARY OUTCOMES:
Effect of Lapband-induced weight loss on quality of life | 18 months
  Measured using the Expanded Prostate Cancer Index Composite (EPIC). The EPIC for Clinical Practice (EPIC-CP) is a one-page, 16-item questionnaire to measure urinary incontinence, urinary irritation, bowel, sexual, and hormonal HRQOL domains
Effect of Lapband-induced weight loss on sexual function | 18 months
  Measured using EPIC and Sexual Health Inventory for Men (SHIM)
Effect of Lapband-induced weight loss on prostate size and associated urinary symptoms | 18 months
  Measured using EPIC and the International Prostate Symptom Score (IPSS)
Receiver Operating Curve (ROC) analysis to evaluate PSA cancer detection performance | 18 months
  ROC analysis - prostate cancer vs. no prostate cancer (1-specificity vs. sensitivity for all cutoff values in the range of all PSA levels observed)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wynberg, MD, Principal Investigator — MMC
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States